CLINICAL TRIAL: NCT01908543
Title: Iron Deficiency and Hereditary Haemorrhagic Telangiectasia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical issues with availability of relevant personnel
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLS 2013/1
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Hereditary Haemorrhagic Telangiectasia
Keywords: Iron deficiency; Nosebleeds
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Iron Deficiencies; Epistaxis | interventions — ferrous sulfate; Tablets; Iron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Iron treatment (Experimental): INTERVENTION: Ferrous sulphate 200mg oral tablet
  This is a single arm study. Individuals in this arm will
  * have an additional 15 mls of supplementary research bloods taken with their usual clinic bloods
  * receive a single tablet of ferrous sulphate 200mg
  * fill in questionnaires that formally evaluate their nosebleed losses and dietary iron intake in the preceding 12 months
  * have a second blood sample later that day (20 mls of blood
  Total number of participants in arm = 100
  Interventions: Drug: Ferrous sulphate 200mg oral tablet

INTERVENTIONS:
Drug: Ferrous sulphate 200mg oral tablet — Administration by mouth
  Other Names: Iron tablet

SUMMARY:
Managing iron deficiency is important for more than 1 billion individuals worldwide, to avoid blood transfusions, or excessive strain on vital organs that depend on iron-containing haemoglobin to deliver oxygen to the tissues. Iron deficiency is a particular problem for people with the inherited condition hereditary haemorrhagic telangiectasia (HHT). Their iron deficiency and anaemia results from blood losses, especially from the nose (nosebleeds, and they often need additional iron to replace that lost through bleeding.

Our goal is to stratify HHT patients into high/low absorbers of iron; to define what extra iron they need to adjust for their current and likely future blood losses; and to work out how to achieve this most safely for each individual to improve their later health.

We will test the hypothesis that informed assessment of iron intake and post absorption cellular profiles changes the recommendations for iron intake for HHT patients.

DETAILED DESCRIPTION:
Relevant patients due to come to clinic or the programmed investigation unit will be offered the opportunity to participate in the study.

Up to 100 consenting individuals will

* have an additional 15 mls of supplementary research bloods taken
* receive a single tablet of ferrous sulphate 200mg
* fill in questionnaires that formally evaluate their nosebleed losses and dietary iron intake in the preceding 12 months
* have a second blood sample later that day (20 mls of blood)

The primary outcome measure is the change in serum iron levels post iron tablet.

Other outcome measures will include:

* Haematinic indices indicating whether their iron requirements have been met previously.
* Additional predicted iron intake requirements to adjust for haemorrhagic iron losses

ELIGIBILITY:
Inclusion Criteria:

* Hereditary haemorrhagic telangiectasia (HHT). Definite diagnosis of HHT by international criteria.
* No iron tablets or treatment taken on day of assessment
* Ability to provide informed consent.

Exclusion Criteria:

* Inability to provide informed consent
* Intercurrent infection or illness predicted to modify iron absorption.
* Needle phobia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Blood iron indices | 4-5 hours after iron tablet ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Claire L Shovlin, PhD FRCP, Principal Investigator — Imperial College London
Locations (1):
- Wellcome Trust-McMichael Clinical Research Facility, Imperial college London London, United Kingdom W12 0NN, London, United Kingdom